CLINICAL TRIAL: NCT01294137
Title: Accuracy of Pulse Oximetry to Detect Sleep Apnea in Frail Hospitalized Patients
Brief Title: Sleep Apnea in Frail Elderly
Acronym: SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AGIR à Dom (Other)
Responsible Party: Dr Maziere Sylvie, CHU, Grenoble, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-AGIR-3
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2011-02

CONDITIONS: Ageing; Sleep Apnea
Keywords: frail; elderly; hospitalized; sleep apnea; oximetry
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ventilatory polygraphy (Active Comparator)
  Interventions: Device: ventilatory polygraphy

INTERVENTIONS:
Device: ventilatory polygraphy

SUMMARY:
Sleep apnea syndrome is common and increases with age. In the elderly, symptoms might be different than in the youngest people, and its consequences might be severe and atypical (falls, functional and cognitive decline).

Today, there is no specific tool to detect sleep apnea in the elderly. The goal of this study is to evaluate the accuracy of oximetry for detection of respiratory disturbances in sleep apnea in the hospitalized elderly.

DETAILED DESCRIPTION:
Main goal: to define the more specific and sensitive cut-off of variability index of the oximetry to detect sleep apnea in the hospitalized elderly.

Secondary goals:

* sleep apnea prevalence in the elderly
* accuracy of other oximetry parameters (saturation line, oximetry desaturation index, autonomic arousals) for detection of respiratory disturbances in sleep apnea in the hospitalized elderly
* to determine the clinical and biological data associated with sleep apnea in the hospitalized elderly
* to determine the factors associated with the record failures and its prevalence
* to study the prevalence of the Periodic Limb Movements of Sleep in the hospitalized elderly

Study design: simultaneous records by oximetry and ventilatory polygraphy with tibial EMG in the hospitalized elderly in a geriatric readaptation unit.

ELIGIBILITY:
Inclusion Criteria:

* age > 75 ans
* affiliation to the French health care system

Exclusion Criteria:

* hypoxemia with oxygenotherapy
* already known and treated sleep apnea syndrome
* mild to severe dementia (MMSE<18/30)
* nocturnal neurpsychological disturbances
* acute organic failure

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Maziere, MD, Principal Investigator — University Hospital, Grenoble; Gaëtan Gavazzi, MD PhD, Study Chair — University Hospital, Grenoble; Catherine Bioteau, MD, Study Chair — University Hospital, Grenoble; Pascal Couturier, MD, PhD, Study Chair — University Hospital, Grenoble; Renaud Tamisier, MD, Study Chair — University Hospital, Grenoble; Sandrine Launois, MD, Study Chair — University Hospital, Grenoble; Patrick Lévy, MD, PhD, Study Chair — University Hospital, Grenoble; Jean-Louis Pépin, MD, PhD, Study Director — University Hospital, Grenoble
Locations (1):
- CHU Grenoble, La Tronche, France